CLINICAL TRIAL: NCT02351414
Title: Post Market Clinical Follow-Up Study of the EVOLUTION® Total Knee Arthroplasty System With Cruciate Sacrificing Inserts
Brief Title: Post Market Follow-Up Study of the EVOLUTION® Total Knee Arthroplasty System With Cruciate Sacrificing Inserts
Acronym: AMETHYST
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-LJK-001
Record Dates: First submitted 2015-01-22; First posted 2015-01-30 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Joint Disease
Keywords: Osteoarthritis; Ankylosis; Revision procedures; Correction of functional deformity; Rheumatoid arthritis; Arthritis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Ankylosis; Arthritis, Rheumatoid; Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Total Knee Arthroplasty: Single study group previously implanted with the EVOLUTION® TKA System with cruciate sacrificing (CS) inserts
  Interventions: Device: Total Knee Arthroplasty (EVOLUTION®)

INTERVENTIONS:
Device: Total Knee Arthroplasty (EVOLUTION®)
  Other Names: EVOLUTION® Total Knee Arthroplasty System with CS Inserts; EVOLUTION® CS

SUMMARY:
MPO is conducting this PMCF study to evaluate the safety and efficacy of its EVOLUTION® Total Knee Arthroplasty (TKA) components marketed in the EU. These types of studies are required by regulatory authorities for all devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with MEDDEV 2.12/2 rev 2.

DETAILED DESCRIPTION:
MicroPort Orthopedics Inc. (MPO) currently markets the EVOLUTION® TKA System globally, including in the European Union (EU). As part of the process for gaining approval to market in the EU, MicroPort is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of this system. These types of studies are required by regulatory authorities for all TKA devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. The objectives of this study are to evaluate component survivorship, cumulative revision rate, functional outcome scores, and subject satisfaction at early, midterm, and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, subjects must meet all of the following criteria:

* Has previously undergone primary TKA for any of the following:
* non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, or avascular necrosis;
* inflammatory degenerative joint disease including rheumatoid arthritis
* correction of functional deformity.
* Subject was implanted with the specified combination of components
* Subject is willing and able to complete required study visits and assessments
* Subject plans to be available through the 10 year postoperative follow-up visit
* Subject is willing to sign the approved Informed Consent document
* Subject must be at least 2 years post TKA prior to informed consent.

Previously implanted bilateral subjects can have both TKAs enrolled in the study provided: 1) the specified combination of components were implanted in both, 2) all other aspects of the Inclusion/Exclusion Criteria are satisfied, 3) enrollment does not exceed the subject count specified in the Clinical Trial Agreement, and 4) the subject agrees to a second Informed Consent document specific to the second TKA. Prospective enrollment of a previously unimplanted knee is not permitted in this study.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* Subject was skeletally immature (less than 21 years of age) at time of implantation
* Subject is currently enrolled in another clinical investigation
* Subject is unwilling or unable to sign the Informed Consent document
* Subject has documented substance abuse issues
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
* Subject has a body mass index (BMI) of greater than 40
* Subject is currently incarcerated or has impending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with the EVOLUTION® TKA System with cruciate sacrificing (CS) inserts
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary endpoints are analysis of survivorship for all components at each follow-up interval out to 10 years

SECONDARY OUTCOMES:
Patient functional outcomes scores (assessed by KOOS Scores and EQ-5D-3L Scores) | 2-<5 years, 5-7 years, and 10 years
  To characterize functional scores for subjects, as assessed by KOOS Scores and EQ-5D-3L Scores
Cumulative Revision Rate | 2-<5 years, 5-7 years, and 10 years
  To determine the cumulative revision rate at specified intervals out to 10 years follow-up
Subject Satisfaction (assessed by Patient Satisfaction Questionnaires) | 2-<5 years, 5-7 years, and 10 years
  To assess subject satisfaction with their TKA procedure
Number of Radiolucencies | 2-<5 years, 5-7 years, and 10 years
  To summarize the number of radiolucencies in zones surrounding implanted components
Size of Radiolucencies | 2-<5 years, 5-7 years, and 10 years
  To summarize the size of radiolucencies in zones surrounding implanted components

CONTACTS AND LOCATIONS:
Locations (5):
- Illinois Bone & Joint Institute, Morton Grove, Illinois, United States
- AZ Maria-Middelares, Ghent, Belgium
- The Ottawa Hospital, Ottawa, Ontario, Canada
- Klinik für Orthopädie, Unfall- und Wiederherstellungschirurgie, St. Marien Hospital Mülheim an der Ruhr, Mülheim, Germany
- University Hospital Llandough, Penarth, South Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No